CLINICAL TRIAL: NCT00913393
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study of FG-3019 in Subjects With Type 2 Diabetes Mellitus (DM) and Persistent Proteinuria on Background Angiotensin Converting Enzyme Inhibitor (ACEi) and/or Angiotensin II Receptor Blockade (ARB) Therapy
Brief Title: Study of FibroGen (FG)-3019 in Subjects With Type 2 Diabetes Mellitus and Kidney Disease on ACEi and/or ARB Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early for business purposes and as a result of a strategic decision to shift focus to another indication.
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FGCL-3019-032
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Nephropathy; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — pamrevlumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo IV
  Interventions: Drug: Placebo
- 2 (Experimental): 3 mg/kg FG-3019 IV
  Interventions: Drug: FG-3019
- 3 (Experimental): 10 mg/kg FG-3019 IV
  Interventions: Drug: FG-3019

INTERVENTIONS:
Drug: FG-3019 — 3 mg/kg FG-3019 IV every 2 weeks for 22 weeks
  Arms: 2
Drug: FG-3019 — 10 mg/kg FG-3019 IV every 2 weeks for 22 weeks
  Arms: 3
Drug: Placebo — Placebo IV every 2 weeks for 22 weeks
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the effect of FG-3019 on diabetic kidney disease or diabetic nephropathy.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effect of FG-3019 on proteinuria as assessed by urinary albumin/creatinine ratio (ACR).

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed written informed consent
2. Males and females 18-75 years of age, inclusive
3. Diagnosis of type 2 diabetes mellitus according to American Diabetes Association (ADA) criteria
4. 24-hour urinary ACR 200-3000 mg/g, inclusive, on two occasions during screening at least 2 days apart
5. Estimated glomerular filtration rate (eGFR) (by MDRD equation) >20 mL/min/1.73 m2
6. Mean systolic blood pressure less than or equal to 150 mmHg and a mean diastolic blood pressure less than or equal to 95 mmHg
7. Receiving ACEi and/or ARB therapy at an unchanged dose at or above the minimum trial dosage for at least 3 months prior to the first Screening visit and willing to maintain these doses throughout the treatment period

Key Exclusion Criteria:

1. Females who are pregnant or breast feeding
2. Organ transplant recipient, history of dialysis, or known non-diabetic renal disease other than benign cysts or anatomical variants
3. History of New York Heart Association class III/IV heart failure
4. Screening electrocardiogram showing acute and/or clinically significant findings including but not limited to ST depression
5. History of any of the following events within 3 months prior to Screening: coronary artery bypass graft, cerebrovascular accident, myocardial infarction, transient ischemic attack, unstable angina, uncontrolled cardiac arrhythmia, atrial fibrillation, percutaneous coronary intervention, or vascular stent placement
6. History of anaphylactic or systemic allergic reaction to human, humanized, chimeric, or murine monoclonal antibodies
7. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 times the upper limit of normal; direct bilirubin above the upper limit of normal, or >2.5 times the upper limit of normal in cases of documented Gilbert's syndrome
8. Hemoglobin <10 g/dL
9. Hemoglobin A1c (HbA1c) >9 %
10. Low density lipoprotein (LDL) >130 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Measure: change from baseline in 24-hour urinary ACR for each arm compared with placebo | 6 months

SECONDARY OUTCOMES:
Measure: Safety and tolerability of FG-3019 in the study population. | 12 months
Measure: Change from baseline in eGFR for each FG-3019 arm compared to placebo | 6 months
Measure: Change from baseline in serum creatinine for each FG-3019 arm compared with placebo | 6 months

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Tempe, Arizona
  - Buena Park, California
  - Lakewood, California
  - Sacramento, California
  - Walnut Creek, California
  - Whittier, California
  - Atlanta, Georgia
  - Evergreen Park, Illinois
  - Topeka, Kansas
  - Wichita, Kansas
  - Kenner, Louisiana
  - Springfield, Massachusetts
  - Saint Clair Shores, Michigan
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Buffalo, New York
  - Flushing, New York
  - New York, New York
  - Greenville, North Carolina
  - Toledo, Ohio
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Spokane, Washington